CLINICAL TRIAL: NCT04728828
Title: Immune Response After COVID19 Vaccination in a Multicenter Cohort of In-center Haemodialysis Patients in France
Brief Title: COVADIAL - Immunogenicity of COVID-19 Vaccine in Hemodialysis Patients
Acronym: COVADIAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cornouaille (Other)
Collaborators: Centre Hospitalier Régional et Universitaire de Brest (Other)
Responsible Party: Sponsor
Other Study IDs: COVADIAL
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Covid19
Keywords: Covid19; Vaccine response; Serology; haemodialysis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In-center adult haemodialysis patients eligible and voluntary for COVID19 vaccination
  Interventions: Biological: Serological COVID-19 vaccine immunogenicity

INTERVENTIONS:
Biological: Serological COVID-19 vaccine immunogenicity — Serological test

SUMMARY:
COVID-19 is a severe disease with poor prognosis in patients receiving in-center haemodialysis (HD). A population-based registry of >4,000 patients with a diagnosis of COVID-19 receiving kidney replacement therapy (either haemodialysis or kidney transplant recipient) highlighted a 21.1 fold higher 28-day mortality risk among patients on dialysis (n = 3,285), than the expected 1.2% mortality of propensity-score matched historical controls. Vulnerability in uraemic patients is a combination of intrinsic frailty, increased risk of infection and a high burden of comorbidities. In patients on HD, abnormalities in the immune response may contribute to relative hyporesponsiveness to vaccines. However, patients on HD appear to seroconvert at a similar rate compared to the general population after SARS-CoV-2 infection, suggesting a likelihood of vaccine efficacy but this population has been excluded from vaccine trials. The primary aim of this study is to evaluate antibody synthesis induced after Covid-19 vaccination in a French adult multicentric cohort of in-center haemodialysis patients. The second aim of this study is to identify vaccine non-responders among HD patients and to assess the clinical and biological risk factors associated with non-response.

DETAILED DESCRIPTION:
Hemodialysis patients were excluded from COVID19 vaccine response studies: seroprotection rate? Long-term protection? Different regimens to offer to hemodialysis patients?

ELIGIBILITY:
Inclusion Criteria:

* all in-center haemodialysis individuals eligible and voluntary to receive one of the approved COVID-19 vaccines.

Exclusion Criteria:

* individuals under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all in-center haemodialysis patients eligible to receive one of the approved SARS-CoV-2/COVID-19 vaccines.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
antibody synthesis induced after Covid-19 vaccination (positive or negative) | 1 month after 2nd injection
  evaluation of IgG anti-S level

SECONDARY OUTCOMES:
Lack of immunogenicity | day 0, before 2nd injection, 1 month after reinjection, 3 months after reinjection, 6 months, 12 months, 24 months
  evaluation of IgG anti-S level
COVID-19 incidence | day 0, before 2nd injection, 1 month after reinjection, 3 months after reinjection, 6 months, 12 months, 24 months
Death during follow up | day 0, before 2nd injection, 1 month after reinjection, 3 months after reinjection, 6 months, 12 months, 24 months
measure antibody response to vaccines in patient subgroup (diabetic patients, patients with auto-immune disease, patients with cancer, patients with an history of solid organ transplantation) | day 0, before 2nd injection, 1 month after reinjection, 3 months after reinjection, 6 months, 12 months, 24 months
  evaluation of IgG anti-S level
Longevity of the antibody synthesis induced after Covid-19 vaccination | 3 months after reinjection, 6 months after reinjection, 12 months after reinjection, 24 months after reinjection
  evaluation of IgG anti-S level
antibody synthesis induced after one injection of Covid-19 vaccine | before second injection
  evaluation of IgG anti-S level

OTHER OUTCOMES:
Hepatitis B-vaccination response | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Quimper, Quimper, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jager KJ, Kramer A, Chesnaye NC, Couchoud C, Sanchez-Alvarez JE, Garneata L, Collart F, Hemmelder MH, Ambuhl P, Kerschbaum J, Legeai C, Del Pino Y Pino MD, Mircescu G, Mazzoleni L, Hoekstra T, Winzeler R, Mayer G, Stel VS, Wanner C, Zoccali C, Massy ZA. Results from the ERA-EDTA Registry indicate a high mortality due to COVID-19 in dialysis patients and kidney transplant recipients across Europe. Kidney Int. 2020 Dec;98(6):1540-1548. doi: 10.1016/j.kint.2020.09.006. Epub 2020 Oct 15. PMID 32979369
- [Result] ERA-EDTA Council; ERACODA Working Group. Chronic kidney disease is a key risk factor for severe COVID-19: a call to action by the ERA-EDTA. Nephrol Dial Transplant. 2021 Jan 1;36(1):87-94. doi: 10.1093/ndt/gfaa314. PMID 33340043
- [Result] Eleftheriadis T, Antoniadi G, Liakopoulos V, Kartsios C, Stefanidis I. Disturbances of acquired immunity in hemodialysis patients. Semin Dial. 2007 Sep-Oct;20(5):440-51. doi: 10.1111/j.1525-139X.2007.00283.x. PMID 17897251
- [Result] Mahalingasivam V, Tomlinson L. The seroprevalence of SARS-CoV-2 in patients on haemodialysis. Nat Rev Nephrol. 2021 Apr;17(4):225-226. doi: 10.1038/s41581-020-00379-y. PMID 33230249